CLINICAL TRIAL: NCT00621621
Title: CryoCath Freezor CryoAblation Catheter System (CRYOFACTS)
Acronym: PS-010
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-010
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Tachycardia, Atrioventricular Nodal Reentry
Keywords: atrioventricular nodal reentrant tachycardia; AVNRT
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Freezor Catheter for AVNRT (Experimental): Subjects with Atrio Ventricular Reentrant Tachycardia (AVNRT)will be treated with cryo (freezing) energy to ablate the slow pathway causing the arrythmia.
  Interventions: Device: Freezor® Cardiac Cryoablation Catheter CryoConsole System
- External Data Supporting the Study (Other): This arm was taken from pier reviewed published reports that include adult subjects ablated with the Freezor catheter for AVNRT.
  Interventions: Device: Freezor® Cardiac Cryoablation Catheter CryoConsole System

INTERVENTIONS:
Device: Freezor® Cardiac Cryoablation Catheter CryoConsole System — cryoablation
  Other Names: 7F Freezor Cardiac CryoAblation Catheter

SUMMARY:
The purpose of this post approval study of heart block is to gather additional information regarding how often patients develop heart block (atrioventricular block) after having standard ablation procedure using cryotherapy with the Freezor™ catheter.

DETAILED DESCRIPTION:
Due to the lack of enrollments for the trial. The FDA and Medtronic discussed the inclusion of data found from from published literature (external studies) to corroborate study endpoint. The FDA allowed this data and the study was closed.

ELIGIBILITY:
Inclusion Criteria:

Some inclusion criteria can only be established during the electrophysiologic study (EPS); thus there are two groups of inclusion criteria.

For inclusion in the study subjects must fulfill ALL of the following criteria:

Pre-EPS inclusion criteria:

1. Patients with a clinical history of AVNRT who are referred for ablation.
2. Patients willing to provide written informed consent.

Post-EPS inclusion criteria:

1. Patients with EPS-documented AVNRT

Exclusion Criteria:

ANY of the following is regarded as a criterion for excluding a subject from the study:

1. Patients with any pre-existing AV block.
2. Patients with known cryoglobulinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lehmann, MD, MPH, Principal Investigator — Lehmann Consulting
Locations (4):
- United States (4):
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Medical Center and the New York Presbyterian Hospital, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Background] Friedman PL, Dubuc M, Green MS, Jackman WM, Keane DT, Marinchak RA, Nazari J, Packer DL, Skanes A, Steinberg JS, Stevenson WG, Tchou PJ, Wilber DJ, Worley SJ. Catheter cryoablation of supraventricular tachycardia: results of the multicenter prospective "frosty" trial. Heart Rhythm. 2004 Jul;1(2):129-38. doi: 10.1016/j.hrthm.2004.02.022. PMID 15851143

RESULTS

PARTICIPANT FLOW:
Groups:
- Focal Cryoablation Group: Subjects with Atrio Ventricular Reentrant Tachycardia (AVNRT)will be treated with cryo (freezing) energy to ablate the slow pathway causing the arrythmia.
  Freezor® Cardiac Cryoablation Catheter CryoConsole System: cryoablation
- External Data Supporting the Study: Data from published reports that include subjects that met inclusion criteria for study and contained data of Heart block.
Period: Overall Study
Arm/Group | Focal Cryoablation Group | External Data Supporting the Study
Started | 105 (Date of Post- Approval Study protocol approval) | 705
Completed | 75 (Treated with the experimental catheter) | 705
Not Completed | 30 | 0
Not completed — Subjects were exited at EP study | 30 | 0

BASELINE CHARACTERISTICS:
Population: A total of 105 subjects gave actual consent in the study. Of the 105 consented 75 went on to have an ablation procedure performed. Data from 675 subjects were taken from published data that met inclusion criteria with publication search approved by the FDA.
Groups:
- Subjects Consented in the Study Not Ablated: Actual Subjects that were consented in the study that did not meet inclusion criteria.
- Subjects Collected From Published Data: Published evidence about the safety and efficacy of using Medtronic's Freezor® 4 mm CryoCatheter has been reported since the initiation of the CryoFACTS-PAS. The results reported in the literature provide the supplemental data in the same study population as in the PAS and are included to meet the study objectives, as agreed upon with the FDA.
- Total: Total of all reporting groups
Arm/Group | Focal Cryoablation Group | Subjects Consented in the Study Not Ablated | Subjects Collected From Published Data | Total
Number analyzed (Participants) | 75 | 30 | 675 | 780
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (17.8) | NA (NA) — Data was not collected on subjects that were not ablated by the site. | NA (NA) — Data was not collected on subjects that were not ablated by the site. | NA (NA) — Data was not collected on subjects that were not ablated by the site.
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline demographics were only collected for actual enrolled subjects (n=75) That were ablated. This data was not available for subjects enrolled from publicaton data (675).
  Participants
    Female | 55 | NA — Data was not collected on subjects that were not ablated by the site. | NA — Data was not collected on subjects that were not ablated by the site. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | 20 | NA — Data was not collected on subjects that were not ablated by the site. | NA — Data was not collected on subjects that were not ablated by the site. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 75 | 30 | NA — Regions were not collected from Publication data | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Device or Procedure Related AV Block Persistent Through Discharge From Hospital.
Time Frame: After 250 subjects have been enrolled.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Focal Cryoablation Group | External Data Supporting the Study
Number analyzed (Participants) | 75 | 705
participants | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]

2. Secondary Outcome: AV Block That Requires the Insertion of a Permanent Pacemaker: Defined as the Insertion of a Permanent Pacemaker, as Assessed During Defined Study Follow up.
Time Frame: After 250 subjects have been enrolled.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Experimental: Freezor Catheter for AVNRT: Subjects with Atrio Ventricular Reentrant Tachycardia (AVNRT)will be treated with cryo (freezing) energy to ablate the slow pathway causing the arrythmiacryoablation
Arm/Group | Experimental: Freezor Catheter for AVNRT | External Data Supporting the Study
Number analyzed (Participants) | 75 | 705
participants | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]

ADVERSE EVENTS:
Groups:
- External Data Supporting the Study: Subjects from publication search with Atrio Ventricular Reentrant Tachycardia (AVNRT)will be treated with cryo (freezing) energy to ablate the slow pathway causing the arrythmia.
  Freezor® Cardiac Cryoablation Catheter CryoConsole System: cryoablation
Arm/Group | Focal Cryoablation Group | External Data Supporting the Study
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/705
Other Adverse Events (participants affected / at risk) | 0/75 | 0/705

LIMITATIONS AND CAVEATS:
Slow enrollment in the trial showed limited the amount of available data. Detailed subject data from the published literature was not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less